CLINICAL TRIAL: NCT01000727
Title: A Clinical Outcomes Study of Darapladib Versus Placebo in Subjects Following Acute Coronary Syndrome to Compare the Incidence of Major Adverse Cardiovascular Events (MACE).
Brief Title: The Stabilization Of pLaques usIng Darapladib-Thrombolysis In Myocardial Infarction 52 Trial
Acronym: SOLID-TIMI 52
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: The TIMI Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 480848/033
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Results first posted 2017-08-10 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-06

CONDITIONS: Acute Coronary Syndrome
Keywords: Atherosclerosis; Heart disease; Cardiovascular disease; Lp-PLA2 inhibitor; The TIMI Study Group; Coronary Heart Disease (CHD); Acute Coronary Syndrome (ACS)
MeSH Terms: conditions — Acute Coronary Syndrome; Atherosclerosis; Heart Diseases; Cardiovascular Diseases; Coronary Disease | interventions — darapladib; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Darapladib 160 mg (Experimental): Single daily oral tablet
  Interventions: Drug: Darapladib 160 mg; Other: Standard Therapy
- Placebo (Placebo Comparator): Single daily oral tablet
  Interventions: Drug: Placebo; Other: Standard Therapy

INTERVENTIONS:
Drug: Darapladib 160 mg — Lp-PLA2 inhibitor
  Other Names: SB-480848
  Arms: Darapladib 160 mg
Drug: Placebo — Placebo administered
  Arms: Placebo
Other: Standard Therapy — Guideline mandated therapy for individual's condition

SUMMARY:
This study will test whether darapladib can safely lower the chances of having a cardiovascular event (such as a heart attack or urgent coronary revascularization (e.g. medical procedures performed to restore the normal blood flow in patients with atherosclerosis)) when treatment is started within 30 days after an acute coronary syndrome (also called ACS).

DETAILED DESCRIPTION:
Subjects who qualify for the study will be randomized 1:1 to either darapladib or placebo administered in addition to standard therapy. Following the baseline visit, subjects will be expected to return for clinic visits at 1 month, 3 months, 6 months and every 6 months until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Men or women at least 18 years old (in Taiwan, at least 20 years old). Women must be post-menopausal or using a highly effective method for avoidance of pregnancy.
* Hospitalization for acute coronary syndrome (ACS) within 30 days prior to study entry.
* Clinically stable for 24 hours prior to study entry.
* A planned percutaneous coronary intervention (PCI) should be performed prior to study entry, whenever possible.
* At least one of the following:
* At least 60 years old.
* Myocardial infarction prior to the qualifying ACS event.
* Diabetes mellitus requiring treatment with medication.
* Diagnosed mild or moderate reduction in kidney function.
* Cerebrovascular disease (carotid artery disease or ischemic stroke more than 3 months prior to study entry) OR peripheral artery disease.

Exclusion Criteria:

* ACS symptoms or lab results not believed to be caused by a narrowing or blocked coronary artery.
* No major coronary artery with a blockage of more than 50% (unless all stenoses are successfully treated by PCI).
* Planned coronary artery bypass graft (CABG) surgery, or CABG surgery performed after the qualifying ACS event and prior to study entry.
* Certain types of liver disease.
* Severe reduction in kidney function OR removal of a kidney OR kidney transplant.
* Severe heart failure.
* Blood pressure higher than normal despite lifestyle changes and treatment with medications.
* Any life-threatening disease with a life expectancy of less than 2 years (other than heart disease) that may prevent the subject from completing the study.
* Severe asthma that is poorly controlled with medication.
* Pregnancy (Note: A pregnancy test will be performed on all non-sterile women prior to study entry).
* Previous severe allergic reaction to food, medications, drink, insect stings, etc.
* Drug or alcohol abuse within the past 6 months. Mental/psychological impairment that may prevent the subject from complying with study procedures or understanding the goal and potential risks of participating in the study.
* Certain medications that may interfere with the study medication (these will be identified by the study doctor).
* If both birth parents are at least 50% Japanese, Chinese, or Korean ancestry, must have a blood sample collected for Lp-PLA2 activity. Those with Lp-PLA2 activity less than or equal to 20.0 nmol/min/mL are excluded.
* Previously took darapladib (SB-480848).
* Participation in a study of an investigational medication within the past 30 days.
* Current participation in a study of an investigational device.
* Any other reason the investigator deems the subject should not participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13026 (Actual)
Dates: Start 2009-12-01; Primary Completion 2014-04-01 (Actual); Study Completion 2014-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (719):
- United States (255):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Anchorage, Alaska
  - GSK Investigational Site, Cottonwood, Arizona
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Fort Smith, Arkansas
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Glendale, California
  - GSK Investigational Site, La Mesa, California
  - GSK Investigational Site, Lomita, California
  - GSK Investigational Site, Los Alamitos, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Mission Hills, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Santa Ana, California
  - GSK Investigational Site, Stockton, California
  - GSK Investigational Site, Thousand Oaks, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Ventura, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Golden, Colorado
  - GSK Investigational Site, Greeley, Colorado
  - GSK Investigational Site, Littleton, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Bridgeport, Connecticut
  - GSK Investigational Site, Guilford, Connecticut
  - GSK Investigational Site, Hartford, Connecticut
  - GSK Investigational Site, Atlantis, Florida
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Brandon, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Daytona Beach, Florida
  - GSK Investigational Site, Fleming Island, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Gulf Breeze, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Inverness, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Jacksonville Beach, Florida
  - GSK Investigational Site, Jupiter, Florida
  - GSK Investigational Site, Kissimmee, Florida
  - GSK Investigational Site, Miramar, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Palm Beach Gardens, Florida
  - GSK Investigational Site, Pensacola, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Port Charlotte, Florida
  - GSK Investigational Site, Safety Harbor, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Trinity, Florida
  - GSK Investigational Site, Vero Beach, Florida
  - GSK Investigational Site, Wellington, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Cumming, Georgia
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Aurora, Illinois
  - GSK Investigational Site, Bannockburn, Illinois
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Melrose Park, Illinois
  - GSK Investigational Site, Mokena, Illinois
  - GSK Investigational Site, North Chicago, Illinois
  - GSK Investigational Site, Oakbrook Terrace, Illinois
  - GSK Investigational Site, Park Ridge, Illinois
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, Rock Island, Illinois
  - GSK Investigational Site, Avon, Indiana
  - GSK Investigational Site, Fort Wayne, Indiana
  - GSK Investigational Site, Hammond, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Muncie, Indiana
  - GSK Investigational Site, Munster, Indiana
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Valparaiso, Indiana
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, West Des Moines, Iowa
  - GSK Investigational Site, Crestview Hills, Kentucky
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Alexandria, Louisiana
  - GSK Investigational Site, Lafayette, Louisiana
  - GSK Investigational Site, Lake Charles, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Bangor, Maine
  - GSK Investigational Site, Lewiston, Maine
  - GSK Investigational Site, Scarborough, Maine
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Bel Air, Maryland
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Salisbury, Maryland
  - GSK Investigational Site, Towson, Maryland
  - GSK Investigational Site, Ayer, Massachusetts
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Fall River, Massachusetts
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Worcester, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Dearborn, Michigan
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Flint, Michigan
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Marquette, Michigan
  - GSK Investigational Site, Pontiac, Michigan
  - GSK Investigational Site, Troy, Michigan
  - GSK Investigational Site, Ypsilanti, Michigan
  - GSK Investigational Site, Duluth, Minnesota
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Robbinsdale, Minnesota
  - GSK Investigational Site, Saint Cloud, Minnesota
  - GSK Investigational Site, Saint Paul, Minnesota
  - GSK Investigational Site, Tupelo, Mississippi
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, Joplin, Missouri
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Columbia Falls, Montana
  - GSK Investigational Site, Great Falls, Montana
  - GSK Investigational Site, Kalispell, Montana
  - GSK Investigational Site, Grand Island, Nebraska
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Papillion, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Browns Mills, New Jersey
  - GSK Investigational Site, Elizabeth, New Jersey
  - GSK Investigational Site, Elmer, New Jersey
  - GSK Investigational Site, Haddon Heights, New Jersey
  - GSK Investigational Site, Linden, New Jersey
  - GSK Investigational Site, Paterson, New Jersey
  - GSK Investigational Site, Pomona, New Jersey
  - GSK Investigational Site, Sewell, New Jersey
  - GSK Investigational Site, Somerset, New Jersey
  - GSK Investigational Site, Summit, New Jersey
  - GSK Investigational Site, Voorhees Township, New Jersey
  - GSK Investigational Site, West Orange, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Peekskill, New York
  - GSK Investigational Site, Roslyn, New York
  - GSK Investigational Site, Stony Brook, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Troy, New York
  - GSK Investigational Site, Williamsville, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Burlington, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Concord, North Carolina
  - GSK Investigational Site, Gastonia, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Huntersville, North Carolina
  - GSK Investigational Site, Matthews, North Carolina
  - GSK Investigational Site, Monroe, North Carolina
  - GSK Investigational Site, Pinehurst, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Rocky Mount, North Carolina
  - GSK Investigational Site, Salisbury, North Carolina
  - GSK Investigational Site, Sanford, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Grand Forks, North Dakota
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Elyria, Ohio
  - GSK Investigational Site, Fairfield, Ohio
  - GSK Investigational Site, Fairview Park, Ohio
  - GSK Investigational Site, Lorain, Ohio
  - GSK Investigational Site, Mansfield, Ohio
  - GSK Investigational Site, Middleburg Heights, Ohio
  - GSK Investigational Site, Oakbrook Terrace, Ohio
  - GSK Investigational Site, Sandusky, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Youngstown, Ohio
  - GSK Investigational Site, Zanesville, Ohio
  - GSK Investigational Site, Midwest City, Oklahoma
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Allentown, Pennsylvania
  - GSK Investigational Site, Beaver, Pennsylvania
  - GSK Investigational Site, Bethlehem, Pennsylvania
  - GSK Investigational Site, Camp Hill, Pennsylvania
  - GSK Investigational Site, Chambersburg, Pennsylvania
  - GSK Investigational Site, Doylestown, Pennsylvania
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, Jenkintown, Pennsylvania
  - GSK Investigational Site, Jersey Shore, Pennsylvania
  - GSK Investigational Site, Lancaster, Pennsylvania
  - GSK Investigational Site, Lansdale, Pennsylvania
  - GSK Investigational Site, Leetsdale, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Sayre, Pennsylvania
  - GSK Investigational Site, Scranton, Pennsylvania
  - GSK Investigational Site, Sellersville, Pennsylvania
  - GSK Investigational Site, West Chester, Pennsylvania
  - GSK Investigational Site, York, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Rapid City, South Dakota
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Columbia, Tennessee
  - GSK Investigational Site, Jackson, Tennessee
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Oak Ridge, Tennessee
  - GSK Investigational Site, Amarillo, Texas
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Galveston, Texas
  - GSK Investigational Site, Harker Heights, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Katy, Texas
  - GSK Investigational Site, Kingwood, Texas
  - GSK Investigational Site, Round Rock, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, San Marcos, Texas
  - GSK Investigational Site, Sugar Land, Texas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Victoria, Texas
  - GSK Investigational Site, Lynchburg, Virginia
  - GSK Investigational Site, Midlothian, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Winchester, Virginia
  - GSK Investigational Site, Bellevue, Washington
  - GSK Investigational Site, Bellingham, Washington
  - GSK Investigational Site, Burien, Washington
  - GSK Investigational Site, Everett, Washington
  - GSK Investigational Site, Kirkland, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Walla Walla, Washington
  - GSK Investigational Site, Beloit, Wisconsin
  - GSK Investigational Site, Green Bay, Wisconsin
  - GSK Investigational Site, Madison, Wisconsin
  - GSK Investigational Site, Wausau, Wisconsin
- Argentina (16):
  - GSK Investigational Site, Capital Federal, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, Ramos Mejía, Buenos Aires
  - GSK Investigational Site, San Justo, Buenos Aires
  - GSK Investigational Site, San Nicolás de los Arroyos, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Cipolletti
  - GSK Investigational Site, Corrientes
  - GSK Investigational Site, Haedo, Buenos Aires
  - GSK Investigational Site, San Miguel de Tucumán
  - GSK Investigational Site, Santa Fe
  - GSK Investigational Site, Sante Fe
  - GSK Investigational Site, Zárate
- Australia (13):
  - GSK Investigational Site, Garran, Australian Capital Territory
  - GSK Investigational Site, Camperdown, New South Wales
  - GSK Investigational Site, Gosford, New South Wales
  - GSK Investigational Site, Auchenflower, Queensland
  - GSK Investigational Site, Herston, Queensland
  - GSK Investigational Site, Milton, Queensland
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Elizabeth Vale, South Australia
  - GSK Investigational Site, Hobart, Tasmania
  - GSK Investigational Site, Box Hill, Victoria
  - GSK Investigational Site, Nedlands, Victoria
  - GSK Investigational Site, Fremantle, Western Australia
  - GSK Investigational Site, Ashford
- Belgium (9):
  - GSK Investigational Site, Aalst
  - GSK Investigational Site, Bonheiden
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Genk
  - GSK Investigational Site, La Louvière
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Roeselaere
- Brazil (21):
  - GSK Investigational Site, Fortaleza, Ceará
  - GSK Investigational Site, Salvador, Estado de Bahia
  - GSK Investigational Site, Goiânia - GO, Goiás
  - GSK Investigational Site, Belo Horizonte, Minas Gerais
  - GSK Investigational Site, Campina Grande do Sul, Paraná
  - GSK Investigational Site, Curitiba, Paraná
  - GSK Investigational Site, Natal, Rio Grande do Norte
  - GSK Investigational Site, Pelotas, Rio Grande do Sul
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Marília, São Paulo
  - GSK Investigational Site, São José do Rio Preto, São Paulo
  - GSK Investigational Site, São Paulo, São Paulo
  - GSK Investigational Site, Votuporanga, São Paulo
  - GSK Investigational Site, Bahia
  - GSK Investigational Site, Brasília
  - GSK Investigational Site, Campinas
  - GSK Investigational Site, Campo Grande
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, São Paulo
  - GSK Investigational Site, São Paulo - SP
  - GSK Investigational Site, Uberlândia
- Bulgaria (6):
  - GSK Investigational Site, Dimitrovgrad
  - GSK Investigational Site, Haskovo
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Veliko Tarnovo
- Canada (26):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Campbell River, British Columbia
  - GSK Investigational Site, New Westminster, British Columbia
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Ajax, Ontario
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Cambridge, Ontario
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Kelowna, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Newmarket, Ontario
  - GSK Investigational Site, Oshawa, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Sarnia, Ontario
  - GSK Investigational Site, Thunder Bay, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Longueuil, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Thetford-Mines, Quebec
- Chile (7):
  - GSK Investigational Site, Temuco, Región de La Araucania
  - GSK Investigational Site, Viña del Mar, Región de Valparaíso
  - GSK Investigational Site, Concepción, Región Del Biobio
  - GSK Investigational Site, Talcahuano, Región Del Biobio
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago
  - GSK Investigational Site, Temuco
- China (17):
  - GSK Investigational Site, Lanzhou, Gansu
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Nanning, Guangxi
  - GSK Investigational Site, Haikou, Hainan
  - GSK Investigational Site, Shijiazhuang, Hebei
  - GSK Investigational Site, Nanjing, Jiangsu
  - GSK Investigational Site, Dalian, Liaoning
  - GSK Investigational Site, Shenyang, Liaoning
  - GSK Investigational Site, Xi'an, Shaanxi
  - GSK Investigational Site, Jinan, Shandong
  - GSK Investigational Site, Chengdu, Sichuan
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Jinan
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Suzhou
- Colombia (7):
  - GSK Investigational Site, Armenia
  - GSK Investigational Site, Barranquilla
  - GSK Investigational Site, Bogotá
  - GSK Investigational Site, Bucaramanga
  - GSK Investigational Site, Cartagena
  - GSK Investigational Site, Manizales
  - GSK Investigational Site, Medellín
- Czechia (12):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Čáslav
  - GSK Investigational Site, Jihlava
  - GSK Investigational Site, Kroměříž
  - GSK Investigational Site, Milevsko
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Plzen - Bory
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Slaný
  - GSK Investigational Site, Svitavy
  - GSK Investigational Site, Ústí nad Orlicí
  - GSK Investigational Site, Zlín
- Denmark (19):
  - GSK Investigational Site, Aalborg
  - GSK Investigational Site, Aarhus
  - GSK Investigational Site, Esbjerg
  - GSK Investigational Site, Frederikssund
  - GSK Investigational Site, Glostrup Municipality
  - GSK Investigational Site, Hellerup
  - GSK Investigational Site, Herlev
  - GSK Investigational Site, Holbæk
  - GSK Investigational Site, Hvidovre
  - GSK Investigational Site, Koebenhavn N
  - GSK Investigational Site, Kolding
  - GSK Investigational Site, København NV
  - GSK Investigational Site, København S
  - GSK Investigational Site, Køge
  - GSK Investigational Site, Næstved
  - GSK Investigational Site, Odense C
  - GSK Investigational Site, Roskilde
  - GSK Investigational Site, Silkeborg
  - GSK Investigational Site, Svendborg
- France (21):
  - GSK Investigational Site, Pau, Aquitaine
  - GSK Investigational Site, Langres, Champagne-Ardenne
  - GSK Investigational Site, Dunkirk, Hauts-de-France
  - GSK Investigational Site, Avignon
  - GSK Investigational Site, Besançon
  - GSK Investigational Site, Bron
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, Lagny-sur-Marne
  - GSK Investigational Site, Le Plessis-Robinson
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montfermeil
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Poitiers
  - GSK Investigational Site, Quincy-sous-Sénart
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Tourcoing
  - GSK Investigational Site, Valenciennes
- Germany (28):
  - GSK Investigational Site, Bad Krozingen, Baden-Wurttemberg
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Bad Nauheim, Hesse
  - GSK Investigational Site, Darmstadt, Hesse
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Langen, Hesse
  - GSK Investigational Site, Limburg an der Lahn, Hesse
  - GSK Investigational Site, Bad Rothenfelde, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Oldenburg, Lower Saxony
  - GSK Investigational Site, Bielefeld, North Rhine-Westphalia
  - GSK Investigational Site, Eschweiler, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Neuss, North Rhine-Westphalia
  - GSK Investigational Site, Wuppertal, North Rhine-Westphalia
  - GSK Investigational Site, Ludwigshafen am Rhein, Rhineland-Palatinate
  - GSK Investigational Site, Homburg, Saarland
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Altenburg, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Bremen
  - GSK Investigational Site, Halle
  - GSK Investigational Site, Hamburg
- Hungary (11):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Cegléd
  - GSK Investigational Site, Eger
  - GSK Investigational Site, Gyula
  - GSK Investigational Site, Hódmezővásárhely
  - GSK Investigational Site, Kistarcsa
  - GSK Investigational Site, Miskolc
  - GSK Investigational Site, Székesfehérvár
  - GSK Investigational Site, Szolnok
  - GSK Investigational Site, Szombathely
  - GSK Investigational Site, Zalaegerszeg
- India (18):
  - GSK Investigational Site, Ahmedabad
  - GSK Investigational Site, Amritsar
  - GSK Investigational Site, Chennai
  - GSK Investigational Site, Faridabad
  - GSK Investigational Site, Gandhinagar
  - GSK Investigational Site, Gūrgaon
  - GSK Investigational Site, Hyderabad
  - GSK Investigational Site, Indore
  - GSK Investigational Site, Jaipur
  - GSK Investigational Site, Lucknow
  - GSK Investigational Site, Mohali
  - GSK Investigational Site, New Delhi
  - GSK Investigational Site, Noida
  - GSK Investigational Site, Patiāla
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Secunderabad
  - GSK Investigational Site, Vadodara
  - GSK Investigational Site, Visakhapatnam
- Israel (14):
  - GSK Investigational Site, Ashkelon
  - GSK Investigational Site, Beersheba
  - GSK Investigational Site, Haddera
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Holon
  - GSK Investigational Site, Jerusalem
  - GSK Investigational Site, Kfar Saba
  - GSK Investigational Site, Nahariya
  - GSK Investigational Site, Poria – Neve Oved
  - GSK Investigational Site, Raanana
  - GSK Investigational Site, Ramat Gan
  - GSK Investigational Site, Rehovot
  - GSK Investigational Site, Safed
  - GSK Investigational Site, Tel Aviv
- Italy (20):
  - GSK Investigational Site, Catanzaro, Calabria
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Carpi, Emilia-Romagna
  - GSK Investigational Site, Ferrara, Emilia-Romagna
  - GSK Investigational Site, Parma, Emilia-Romagna
  - GSK Investigational Site, Palmanova, Friuli Venezia Giulia
  - GSK Investigational Site, San Daniele del Friuli, Friuli Venezia Giulia
  - GSK Investigational Site, Udine, Friuli Venezia Giulia
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Bergamo, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Rozzano (Mi), Lombardy
  - GSK Investigational Site, Novara, Piedmont
  - GSK Investigational Site, Sassari, Sardinia
  - GSK Investigational Site, Ascoli Piceno, The Marches
  - GSK Investigational Site, Pisa, Tuscany
  - GSK Investigational Site, Treviso, Veneto
  - GSK Investigational Site, Legnano
  - GSK Investigational Site, Sassuolo
- Japan (13):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Ōita
  - GSK Investigational Site, Saga
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
- Netherlands (33):
  - GSK Investigational Site, 's-Hertogenbosch
  - GSK Investigational Site, Amersfoort
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Apeldoorn
  - GSK Investigational Site, Blaricum
  - GSK Investigational Site, Deventer
  - GSK Investigational Site, Dirksland
  - GSK Investigational Site, Doetinchem
  - GSK Investigational Site, Drachten
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Gorinchem
  - GSK Investigational Site, Gouda
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Hardenberg
  - GSK Investigational Site, Harderwijk
  - GSK Investigational Site, Heerenveen
  - GSK Investigational Site, Heerlen
  - GSK Investigational Site, Helmond
  - GSK Investigational Site, Hilversum
  - GSK Investigational Site, Hoofddorp
  - GSK Investigational Site, Hoorn
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, Oss
  - GSK Investigational Site, Roermond
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Sittard-geleen
  - GSK Investigational Site, Sneek
  - GSK Investigational Site, The Hague
  - GSK Investigational Site, Tiel
  - GSK Investigational Site, Tilburg
  - GSK Investigational Site, Veldhoven
  - GSK Investigational Site, Venlo
  - GSK Investigational Site, Zoetermeer
- New Zealand (10):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Dunedin
  - GSK Investigational Site, Hamilton
  - GSK Investigational Site, Lower Hutt
  - GSK Investigational Site, New Plymouth
  - GSK Investigational Site, Palmerston North
  - GSK Investigational Site, Takapuna, Auckland
  - GSK Investigational Site, Tauranga
  - GSK Investigational Site, Whangarei
- Peru (5):
  - GSK Investigational Site, San Martín de Porres, Lima region
  - GSK Investigational Site, Miraflores, Lima, Lima
  - GSK Investigational Site, Callao
  - GSK Investigational Site, Lima
  - GSK Investigational Site, Lima Cercado
- Philippines (4):
  - GSK Investigational Site, Cebu City
  - GSK Investigational Site, Davao City
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Quezon City
- Poland (24):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Bytom
  - GSK Investigational Site, Chrzanów
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Gdynia
  - GSK Investigational Site, Inowrocław
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Lubin
  - GSK Investigational Site, Mielec
  - GSK Investigational Site, Opole
  - GSK Investigational Site, Oława
  - GSK Investigational Site, Radom
  - GSK Investigational Site, Skierniewice
  - GSK Investigational Site, Tarnów
  - GSK Investigational Site, Torun
  - GSK Investigational Site, Tychy
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wałbrzych
  - GSK Investigational Site, Wroclaw
  - GSK Investigational Site, Włocławek
  - GSK Investigational Site, Zamość
  - GSK Investigational Site, Zielona Góra
- Romania (9):
  - GSK Investigational Site, Baia Mare
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Brăila
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Constanța
  - GSK Investigational Site, Craiova
  - GSK Investigational Site, Iași
  - GSK Investigational Site, Târgu Mureş
- Russia (16):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Gatchina
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Krasnoyarsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Orenburg
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, St'Petersburg
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Tyumen
  - GSK Investigational Site, Yaroslavl
  - GSK Investigational Site, Yekaterinburg
- Slovakia (4):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Košice
  - GSK Investigational Site, Nitra
  - GSK Investigational Site, Nové Zámky
- South Africa (15):
  - GSK Investigational Site, Bloemfontein, Free State
  - GSK Investigational Site, Alberton, Gauteng
  - GSK Investigational Site, Johannesburg, Gauteng
  - GSK Investigational Site, Pretoria, Gauteng
  - GSK Investigational Site, Durban, KwaZulu-Natal
  - GSK Investigational Site, Cape Town, Western Province
  - GSK Investigational Site, Panorama, Western Province
  - GSK Investigational Site, Goodwood
  - GSK Investigational Site, Kempton Park
  - GSK Investigational Site, Paarl
  - GSK Investigational Site, Parktown West
  - GSK Investigational Site, Parow
  - GSK Investigational Site, Pretoria
  - GSK Investigational Site, Somerset West
  - GSK Investigational Site, Worcester
- South Korea (7):
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Daejeon
  - GSK Investigational Site, Gangnam-gu, Seoul
  - GSK Investigational Site, Gwangju
  - GSK Investigational Site, Kangwon-do
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seoul
- Spain (13):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, León
  - GSK Investigational Site, Lleida
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Oviedo
  - GSK Investigational Site, San Juan/Alicante
  - GSK Investigational Site, San Sebastián
  - GSK Investigational Site, San Sebastián de Los Reyes/Madrid
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vigo/Pontevedra
- Sweden (7):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Hässleholm
  - GSK Investigational Site, Jönköping
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Östersund
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Västerås
- Taiwan (3):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Yung Kang City
- Thailand (6):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Bangkoknoi
  - GSK Investigational Site, Chiang Mai
  - GSK Investigational Site, Khon Kaen, Muang
  - GSK Investigational Site, Nakhon Ratchasima
  - GSK Investigational Site, Pathum Thani
- Turkey (Türkiye) (4):
  - GSK Investigational Site, Ankara
  - GSK Investigational Site, Erzurum
  - GSK Investigational Site, Eskişehir
  - GSK Investigational Site, Izmir
- Ukraine (11):
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Luhansk
  - GSK Investigational Site, Lutsk
  - GSK Investigational Site, Mykolaiv
  - GSK Investigational Site, Odesa
  - GSK Investigational Site, Simferopol
  - GSK Investigational Site, Vinnytsia
  - GSK Investigational Site, Zaporizhzhya
- United Kingdom (15):
  - GSK Investigational Site, Exeter, Devon
  - GSK Investigational Site, Torquay, Devon
  - GSK Investigational Site, Airdrie, Lanarkshire
  - GSK Investigational Site, Harrow, Middlesex
  - GSK Investigational Site, Northampton, Northamptonshire
  - GSK Investigational Site, Nottingham, Nottinghamshire
  - GSK Investigational Site, Chertsey, Surrey
  - GSK Investigational Site, Coventry, West Midlands
  - GSK Investigational Site, Antrim
  - GSK Investigational Site, Chichester
  - GSK Investigational Site, East Kilbride
  - GSK Investigational Site, Hertfordshire
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, Paisley
  - GSK Investigational Site, Stirling

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Correa S, Morrow DA, Braunwald E, Davies RY, Goodrich EL, Murphy SA, Cannon CP, O'Donoghue ML. Cystatin C for Risk Stratification in Patients After an Acute Coronary Syndrome. J Am Heart Assoc. 2018 Oct 16;7(20):e009077. doi: 10.1161/JAHA.118.009077. PMID 30371283
- [Derived] Barger LK, Rajaratnam SMW, Cannon CP, Lukas MA, Im K, Goodrich EL, Czeisler CA, O'Donoghue ML. Short Sleep Duration, Obstructive Sleep Apnea, Shiftwork, and the Risk of Adverse Cardiovascular Events in Patients After an Acute Coronary Syndrome. J Am Heart Assoc. 2017 Oct 10;6(10):e006959. doi: 10.1161/JAHA.117.006959. PMID 29018021
- [Derived] Eisen A, Cannon CP, Braunwald E, Steen DL, Zhou J, Goodrich EL, Im K, Dalby AJ, Spinar J, Daga S, Lukas MA, O'Donoghue ML. Predictors of Nonuse of a High-Potency Statin After an Acute Coronary Syndrome: Insights From the Stabilization of Plaques Using Darapladib-Thrombolysis in Myocardial Infarction 52 (SOLID-TIMI 52) Trial. J Am Heart Assoc. 2017 Jan 11;6(1):e004332. doi: 10.1161/JAHA.116.004332. PMID 28077384
- [Derived] O'Donoghue ML, Braunwald E, White HD, Lukas MA, Tarka E, Steg PG, Hochman JS, Bode C, Maggioni AP, Im K, Shannon JB, Davies RY, Murphy SA, Crugnale SE, Wiviott SD, Bonaca MP, Watson DF, Weaver WD, Serruys PW, Cannon CP; SOLID-TIMI 52 Investigators; Steen DL. Effect of darapladib on major coronary events after an acute coronary syndrome: the SOLID-TIMI 52 randomized clinical trial. JAMA. 2014 Sep 10;312(10):1006-15. doi: 10.1001/jama.2014.11061. PMID 25173516
- [Derived] O'Donoghue ML, Braunwald E, White HD, Serruys P, Steg PG, Hochman J, Maggioni AP, Bode C, Weaver D, Johnson JL, Cicconetti G, Lukas MA, Tarka E, Cannon CP. Study design and rationale for the Stabilization of pLaques usIng Darapladib-Thrombolysis in Myocardial Infarction (SOLID-TIMI 52) trial in patients after an acute coronary syndrome. Am Heart J. 2011 Oct;162(4):613-619.e1. doi: 10.1016/j.ahj.2011.07.018. Epub 2011 Sep 15. PMID 21982651
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 480848/033 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 480848/033 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 480848/033 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 480848/033 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 480848/033 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 480848/033 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 868 centers in 36 countries: North America (282), Western Europe (210), Eastern Europe (166), Asia/Pacific (127), South America (83) during 07 December 2009 to 24 April 2014. A total of 13026 participants were randomized to the study.
Pre-assignment Details: During the screening phase of the study, participants presenting with acute coronary syndrome (ACS) were randomized within 30 days. Approximately 77% of participants underwent percutaneous coronary intervention (PCI) for the qualifying event.
Groups:
- Placebo: Participants were randomized to receive matching placebo once daily.
- Darapladib 160 mg: Participants were randomized to receive darapladib 160 milligram (mg) enteric-coated tablets once daily.
Period: Overall Study
Arm/Group | Placebo | Darapladib 160 mg
Started | 6522 | 6504
Completed | 6347 | 6328
Not Completed | 175 | 176
Not completed — Lost to Follow-up | 41 | 43
Not completed — Withdrawal by Subject | 111 | 109
Not completed — Study closed/terminated | 23 | 24

BASELINE CHARACTERISTICS:
Groups:
- Darapladib 160 mg: Participants were randomized to receive darapladib 160 mg enteric-coated tablets once daily.
- Total: Total of all reporting groups
Arm/Group | Placebo | Darapladib 160 mg | Total
Number analyzed (Participants) | 6522 | 6504 | 13026
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.3 (9.50) | 64.1 (9.52) | 64.2 (9.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1669 | 1657 | 3326
  Male | 4853 | 4847 | 9700
Race/Ethnicity, Customized [Number; unit: Participants]
  White - White/Caucasian/European Heritage | 5329 | 5331 | 10660
  Asian - East Asian Heritage | 351 | 349 | 700
  Asian - Central/South Asian Heritage | 200 | 211 | 411
  African American/African Heritage | 160 | 155 | 315
  White - Arabic/North African Heritage | 138 | 119 | 257
  Asian - South East Asian Heritage | 123 | 116 | 239
  Asian - Japanese Heritage | 109 | 109 | 218
  American Indian or Alaska Native | 56 | 52 | 108
  Mixed Race | 43 | 52 | 95
  Native Hawaiian or other Pacific Islander | 9 | 5 | 14
  Asian - Mixed Race | 2 | 3 | 5
  White - Mixed Race | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Occurrence of Any Event in the Composite of Major Coronary Events During the Time Period for Follow-up (FU) of Cardiovascular (CV) Event
Description: Coronary heart disease (CHD) death=occurrence of a fatal myocardial infarction (MI), death caused by documented cardiac arrest, death resulting from heart failure in a participant with known CHD, death from other forms of acute/chronic CHD, unwitnessed death of unknown origin, or sudden death. Acute MI=evidence of myocardial necrosis in a clinical setting consistent with myocardial ischemia. Prior MI diagnosed post-randomization (e.g., silent MI)=the development of new pathological Q waves with/without symptoms OR imaging evidence of a region of loss of viable myocardium that is thinned and fails to contract, in the absence of a nonischemic cause (pre-event imaging data required for verification of new abnormality), OR pathological findings of a healed/healing MI. Urgent coronary revascularization (CR) for MI=ischemic discomfort at rest that prompted CR during the same hospitalization or resulted in hospital transfer for the purpose of CR.
Time Frame: From randomization until the End-of-Treatment visit or the last date on which endpoints were able to be assessed (up to 3.80 years)
Population: All-Randomized intent-to-treat (ITT) Population consisted of all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Darapladib 160 mg
Number analyzed (Participants) | 6522 | 6504
Participants | 910 | 903
Statistical Analysis 1: Comparison: Placebo vs Darapladib 160 mg; Test type: Superiority; p = 0.929, Cox Proportional Hazard Regression Model — Statistical significance of this p-value is based on the alpha-spending function of this study; Hazard Ratio (HR) = 1.00, 95.02% CI 2-sided [0.91 to 1.09]

2. Secondary Outcome: Number of Participants With First Occurrence of Any Component of the Composite of Major Adverse Cardiovascular Events (Cardiovascular [CV] Death, Non-fatal MI or Non-fatal Stroke) During the Time Period for Follow-up of CV Events
Description: CV death=death due to a CV cause, which included but was not limited to deaths resulting from stroke, arrhythmia, sudden death (witnessed/unwitnessed), MI, heart failure, pulmonary embolism, peripheral arterial disease, or complications of a CV procedure. Deaths not clearly attributable to non-CV causes are considered to be CV deaths. Acute MI=evidence of myocardial necrosis in a clinical setting consistent with myocardial ischemia. Prior MI diagnosed post-randomization (e.g., silent MI)=the development of new pathological Q waves with/without symptoms OR imaging evidence of a region of loss of viable myocardium that is thinned and fails to contract, in the absence of a non-ischemic cause (pre-event imaging data required for verification of new abnormality), OR pathological findings of a healed/healing MI. Stroke=presence of a new focal neurologic deficit thought to be of vascular origin, with signs/symptoms lasting >24 hours or results in death (in <24 hours).
Time Frame: as for outcome 1
Population: All-Randomized ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Darapladib 160 mg
Number analyzed (Participants) | 6522 | 6504
Participants | 838 | 824
Statistical Analysis 1: Comparison: Placebo vs Darapladib 160 mg; Test type: Superiority; p = 0.777, Cox Proportional Hazard Regression Model — Statistical significance of this p-value is based on the alpha-spending function of this study; Hazard Ratio (HR) = 0.99, 95.02% CI 2-sided [0.90 to 1.09]

3. Secondary Outcome: Number of Participants With Cardiovascular Death During the Time Period for Follow-up of Cardiovascular Events
Description: CV death is defined as a death due to a CV cause, which includes but is not limited to deaths resulting from stroke, arrhythmia, sudden death (witnessed/unwitnessed), MI, heart failure, pulmonary embolism, peripheral arterial disease, or complications of a CV procedure. Deaths not clearly attributable to non-CV causes are considered to be CV deaths.
Time Frame: as for outcome 1
Population: All-Randomized ITT Population
Measure: Count of Participants; unit: Participants
Groups:
- Darapladib 160 mg: Participants were randomized to receive matching placebo once daily.
- Placebo: Participants were randomized to receive darapladib 160 mg enteric-coated tablets once daily.
Arm/Group | Darapladib 160 mg | Placebo
Number analyzed (Participants) | 6522 | 6504
Participants | 268 | 243
Statistical Analysis 1: Comparison: Darapladib 160 mg vs Placebo; Test type: Superiority; p = 0.274, Cox Proportional Hazard Regression Model — Statistical significance of this p-value is based on the alpha-spending function of this study; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.76 to 1.08]

4. Secondary Outcome: Number of Participants With First Occurrence of MI (Fatal/Nonfatal) During the Time Period for Follow-up of Cardiovascular Events
Description: Acute MI is defined as evidence of myocardial necrosis in a clinical setting consistent with myocardial ischemia. Prior MI diagnosed post-randomization (e.g., silent MI)=the development of new pathological Q waves with/without symptoms OR imaging evidence of a region of loss of viable myocardium that is thinned and fails to contract, in the absence of a non-ischemic cause (pre-event imaging data required for verification of new abnormality), OR pathological findings of a healed/healing MI.
Time Frame: as for outcome 1
Population: All-Randomized ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Darapladib 160 mg
Number analyzed (Participants) | 6522 | 6504
Participants | 564 | 547
Statistical Analysis 1: Comparison: Placebo vs Darapladib 160 mg; Test type: Superiority; p = 0.631, Cox Proportional Hazard Regression Model; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.86 to 1.09] — A hazard ratio <1 indicates a lower risk with this treatment compared to Placebo

5. Secondary Outcome: Number of Participants With First Occurrence of Stroke (Fatal/Non-fatal) During the Time Period for Follow-up of Cardiovascular Events
Description: Stroke is defined as the presence of a new focal neurologic deficit thought to be of vascular origin, with signs/symptoms lasting >24 hours or results in death (in <24 hours).
Time Frame: as for outcome 1
Population: All-Randomized ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Darapladib 160 mg
Number analyzed (Participants) | 6522 | 6504
Participants | 130 | 145
Statistical Analysis 1: Comparison: Placebo vs Darapladib 160 mg; Test type: Superiority; p = 0.354, Cox Proportional Hazard Regression Model; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.88 to 1.42] — A hazard ratio < 1 indicates a lower risk with this treatment compared to Placebo

6. Secondary Outcome: Number of Participants With CHD Death During the Time Period for Follow-up of Cardiovascular Events
Description: CHD death is defined as the occurrence of a fatal MI, death caused by documented cardiac arrest, death resulting from heart failure in a participant with known CHD, death from other forms of acute/chronic CHD, unwitnessed death of unknown origin, or sudden death.
Time Frame: as for outcome 1
Population: All-Randomized ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Darapladib 160 mg
Number analyzed (Participants) | 6522 | 6504
Participants | 241 | 211
Statistical Analysis 1: Comparison: Placebo vs Darapladib 160 mg; Test type: Superiority; p = 0.161, Cox Proportional Hazard Regression Model; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.73 to 1.05]

7. Secondary Outcome: Number of Participants With Urgent Coronary Revascularization for Myocardial Ischemia During the Time Period for Follow-up of Cardiovascular Events
Description: Urgent coronary revascularization for myocardial ischemia is defined as ischemic discomfort at rest that prompts coronary revascularization (PCI or coronary artery bypass graft [CABG]) during the same hospitalization or resulting in hospital transfer for the purpose of coronary revascularization. PCI is defined as any attempt at revascularization even if not successful (e.g., angioplasty, atherectomy or stenting).
Time Frame: as for outcome 1
Population: All-Randomized ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Darapladib 160 mg
Number analyzed (Participants) | 6522 | 6504
Participants | 218 | 237
Statistical Analysis 1: Comparison: Placebo vs Darapladib 160 mg; Test type: Superiority; p = 0.360, Cox Proportional Hazard Regression Model; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.91 to 1.31]

8. Secondary Outcome: Number of Participants With First Occurrence of Any Event in the Composite of Total Coronary Events (CHD Death, Non-fatal MI, Hospitalization for Unstable Angina, or Any Coronary Revascularization Procedure) During the Time Period for FU of CV Events
Description: CHD death, acute MI, and prior MI diagnosed post-randomization are defined in the primary endpoint (major coronary events). Hospitalization for unstable angina=one of the following, but not fulfilling the criteria for MI: ischemic discomfort at rest associated with electrocardiogram (ECG) changes leading to hospitalization; ischemic discomfort at rest regardless of ECG changes leading to hospitalization and revascularization during the same admission; ischemic discomfort at rest in hospital associated with ECG changes; ischemic discomfort at rest in hospital without ECG changes resulting in revascularization during the same admission. NOTE: The event was not considered to be unstable angina if, after invasive/non-invasive testing or other diagnostic testing, the discomfort was found not to be caused by myocardial ischemia. Coronary revascularization procedures exclude PCI planned prior to randomization but performed after randomization.
Time Frame: as for outcome 1
Population: All-Randomized ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Darapladib 160 mg
Number analyzed (Participants) | 6522 | 6504
Participants | 1352 | 1290
Statistical Analysis 1: Comparison: Placebo vs Darapladib 160 mg; Test type: Superiority; p = 0.202, Cox Proportional Hazard Regression Model; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.88 to 1.03] — A hazard ratio <1 indicates a lower risk with this treatment compared to Placebo

9. Secondary Outcome: Number of Participants With First Occurrence of Any Coronary Revascularization Procedures (Excluding Coronary Revascularization Planned Prior to Randomization, But Performed After Randomization) During the Time Period for Follow-up of Cardiovascular Event
Description: All coronary revascularization procedures (except for PCI planned prior to randomization but performed after randomization) are included. Examples include coronary artery bypass graft, balloon angioplasty and stenting. The number of participants, with first occurrence of any coronary revascularization procedures, were reported.
Time Frame: as for outcome 1
Population: All-Randomized ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Darapladib 160 mg
Number analyzed (Participants) | 6522 | 6504
Participants | 967 | 926
Statistical Analysis 1: Comparison: Placebo vs Darapladib 160 mg; Test type: Superiority; p = 0.329, Cox Proportional Hazard Regression Model; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.87 to 1.05]

10. Secondary Outcome: Number of Participants With First Occurrence of Any Component of the Composite of All-cause Mortality, Non-fatal MI, or Nonfatal Stroke During the Time Period for Follow-up of Cardiovascular Events
Description: Acute MI is defined as evidence of myocardial necrosis in a clinical setting consistent with myocardial ischemia. Prior MI diagnosed post-randomization (e.g., silent MI)=the development of new pathological Q waves with/without symptoms OR imaging evidence of a region of loss of viable myocardium that is thinned and fails to contract, in the absence of a non-ischemic cause (pre-event imaging data required for verification of new abnormality), OR pathological findings of a healed/healing MI. Stroke=presence of a new focal neurologic deficit thought to be of vascular origin, with signs/symptoms lasting >24 hours or results in death (in <24 hours).
Time Frame: as for outcome 1
Population: All-Randomized ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Darapladib 160 mg
Number analyzed (Participants) | 6522 | 6504
Participants | 928 | 914
Statistical Analysis 1: Comparison: Placebo vs Darapladib 160 mg; Test type: Superiority; p = 0.797, Cox Proportional Hazard Regression Model; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.90 to 1.08]

11. Secondary Outcome: Number of Participants With First Occurrence of Any Event in the Composite of CHD Death and Non-fatal MI During the Time Period for Follow-up of Cardiovascular Events
Description: Acute MI is defined as evidence of myocardial necrosis in a clinical setting consistent with myocardial ischemia. Prior MI diagnosed post-randomization (e.g., silent MI)=the development of new pathological Q waves with/without symptoms OR imaging evidence of a region of loss of viable myocardium that is thinned and fails to contract, in the absence of a non-ischemic cause (pre-event imaging data required for verification of new abnormality), OR pathological findings of a healed/healing MI. CHD death is defined as the occurrence of a fatal MI, death caused by documented cardiac arrest, death resulting from heart failure in a participant with known CHD, death from other forms of acute/chronic CHD, unwitnessed death of unknown origin, or sudden death.
Time Frame: as for outcome 1
Population: All-Randomized ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Darapladib 160 mg
Number analyzed (Participants) | 6522 | 6504
Participants | 725 | 701
Statistical Analysis 1: Comparison: Placebo vs Darapladib 160 mg; Test type: Superiority; p = 0.546, Cox Proportional Hazard Regression Model; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.87 to 1.07] — A hazard ratio <1 indicates a lower risk with this treatment compared to Placebo

12. Secondary Outcome: Number of Participants With All-cause Mortality During the Time Period for Vital Status
Description: Number of participants who died, during the vital status time-period were reported. The participants who were known to have died, date of death was used; for participants who completed the study the study completion date was used; for participants who withdrew from the study where vital status was ascertained , and are known to have not died , the last known date to be alive was used and for participants whom vital status was not ascertained, following study withdrawal the study withdrawal date was used.
Time Frame: as for outcome 1
Population: All-Randomized ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Darapladib 160 mg
Number analyzed (Participants) | 6522 | 6504
Participants | 403 | 376
Statistical Analysis 1: Comparison: Placebo vs Darapladib 160 mg; Test type: Superiority; p = 0.362, Cox Proportional Hazard Regression Model; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.81 to 1.08]

ADVERSE EVENTS:
Time Frame: SAEs and non-serious AEs were collected from start of the study treatment up to 42 days after last dose of study treatment/FU visit.
Description: SAEs and non-serious AEs were collected in members of the Safety Population, comprised of all randomized participants who received at least one dose of investigational product. Post-randomization AEs have an onset date that is on or after the randomization date. The safety population excluded 57 participants in the placebo group and 52 participants in the darapladib group who were randomized but did not receive study drug.
Arm/Group | Placebo | Darapladib 160 mg
All-Cause Mortality (participants affected / at risk) | 403/6465 | 376/6452
Serious Adverse Events (participants affected / at risk) | 3011/6465 | 2933/6452
Other Adverse Events (participants affected / at risk) | 3416/6465 | 3698/6452
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6465) | Darapladib 160 mg (N=6452)
Accelerated hypertension (Vascular disorders) | 1 | 1
Aneurysm (Vascular disorders) | 1 | 1
Angiodysplasia (Vascular disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 11 | 12
Aortic aneurysm rupture (Vascular disorders) | 2 | 0
Aortic dissection (Vascular disorders) | 0 | 1
Aortic occlusion (Vascular disorders) | 1 | 1
Aortic stenosis (Vascular disorders) | 7 | 9
Aortic thrombosis (Vascular disorders) | 0 | 1
Arterial disorder (Vascular disorders) | 1 | 0
Arterial haemorrhage (Vascular disorders) | 1 | 0
Arterial insufficiency (Vascular disorders) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 2 | 0
Arterial thrombosis (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 2 | 3
Arteriovenous fistula (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 1
Coeliac artery occlusion (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 14 | 12
Diabetic microangiopathy (Vascular disorders) | 1 | 1
Embolism (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 4
Femoral artery aneurysm (Vascular disorders) | 1 | 0
Femoral artery dissection (Vascular disorders) | 0 | 1
Femoral artery occlusion (Vascular disorders) | 3 | 3
Haematoma (Vascular disorders) | 4 | 7
Haemodynamic instability (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 38 | 15
Hypertensive crisis (Vascular disorders) | 19 | 13
Hypertensive emergency (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 25 | 18
Hypovolaemic shock (Vascular disorders) | 1 | 0
Iliac artery occlusion (Vascular disorders) | 3 | 6
Iliac artery rupture (Vascular disorders) | 0 | 1
Intermittent claudication (Vascular disorders) | 17 | 15
Ischaemic limb pain (Vascular disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Leriche syndrome (Vascular disorders) | 2 | 1
Lymphatic fistula (Vascular disorders) | 0 | 1
Lymphocele (Vascular disorders) | 1 | 0
Malignant hypertension (Vascular disorders) | 3 | 0
Orthostatic hypotension (Vascular disorders) | 10 | 9
Peripheral arterial occlusive disease (Vascular disorders) | 39 | 36
Peripheral artery aneurysm (Vascular disorders) | 3 | 3
Peripheral artery dissection (Vascular disorders) | 1 | 0
Peripheral artery stenosis (Vascular disorders) | 15 | 25
Peripheral artery thrombosis (Vascular disorders) | 2 | 2
Peripheral embolism (Vascular disorders) | 1 | 2
Peripheral ischaemia (Vascular disorders) | 15 | 17
Peripheral vascular disorder (Vascular disorders) | 15 | 13
Polyarteritis nodosa (Vascular disorders) | 0 | 1
Post thrombotic syndrome (Vascular disorders) | 1 | 0
Reperfusion injury (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 1
Subclavian artery stenosis (Vascular disorders) | 3 | 2
Temporal arteritis (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
Varicose vein (Vascular disorders) | 2 | 2
Vascular insufficiency (Vascular disorders) | 0 | 1
Vascular occlusion (Vascular disorders) | 1 | 1
Vascular pain (Vascular disorders) | 0 | 1
Vascular stenosis (Vascular disorders) | 0 | 1
Vasculitis (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 2
Coronary angioplasty (Surgical and medical procedures) | 1 | 2
Coronary artery bypass (Surgical and medical procedures) | 1 | 2
Percutaneous coronary intervention (Surgical and medical procedures) | 252 | 262
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenosquamous cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Angiocentric lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Angiosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Benign anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 | 10
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2
Bladder cancer stage 0, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bone giant cell tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Borderline ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 10
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Central nervous system neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebellar tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 12
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Cystadenocarcinoma ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Desmoplastic melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 6
Gastric cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Gastrointestinal stromal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glottis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Large cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leiomyosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 12
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 | 11
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung squamous cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 9
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 3
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Metastatic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neurilemmoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Non-small cell lung cancer stage IIIB (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Oral cavity cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Osteosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Paraproteinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pleomorphic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Precursor B-lymphoblastic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 21 | 25
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 7
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 9
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Renal cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Sarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Signet-ring cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Tongue cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tongue carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tonsil cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tracheal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Vaginal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Allergy to arthropod bite (Immune system disorders) | 0 | 1
Allergy to arthropod sting (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 2 | 4
Anaphylactic shock (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 2
Hypersensitivity (Immune system disorders) | 4 | 2
Sarcoidosis (Immune system disorders) | 0 | 1
Asthenia (General disorders) | 4 | 6
Cardiac death (General disorders) | 3 | 2
Chest discomfort (General disorders) | 10 | 8
Chest pain (General disorders) | 15 | 20
Death (General disorders) | 36 | 34
Device dislocation (General disorders) | 1 | 0
Device malfunction (General disorders) | 0 | 3
Device occlusion (General disorders) | 14 | 27
Drug withdrawal syndrome (General disorders) | 0 | 1
Face oedema (General disorders) | 0 | 1
Fatigue (General disorders) | 3 | 1
Gait disturbance (General disorders) | 2 | 1
General physical health deterioration (General disorders) | 2 | 1
Hernia obstructive (General disorders) | 1 | 0
Hypothermia (General disorders) | 1 | 0
Impaired healing (General disorders) | 5 | 1
Inflammation (General disorders) | 1 | 2
Influenza like illness (General disorders) | 0 | 1
Local swelling (General disorders) | 2 | 0
Malaise (General disorders) | 0 | 2
Medical device complication (General disorders) | 1 | 0
Mucosal haemorrhage (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 9 | 3
Nodule (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 298 | 248
Oedema peripheral (General disorders) | 6 | 3
Pain (General disorders) | 0 | 1
Patient-device incompatibility (General disorders) | 1 | 0
Pelvic mass (General disorders) | 1 | 0
Polyserositis (General disorders) | 0 | 1
Pseudopolyp (General disorders) | 0 | 1
Puncture site haemorrhage (General disorders) | 0 | 1
Pyrexia (General disorders) | 11 | 9
Stent malfunction (General disorders) | 0 | 1
Stent-graft endoleak (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 35 | 26
Sudden death (General disorders) | 28 | 26
Surgical failure (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 2
Thrombosis in device (General disorders) | 8 | 8
Ulcer haemorrhage (General disorders) | 1 | 0
Vessel puncture site thrombosis (General disorders) | 1 | 0
Abnormal behaviour (Psychiatric disorders) | 1 | 0
Affective disorder (Psychiatric disorders) | 2 | 0
Alcohol abuse (Psychiatric disorders) | 1 | 2
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0
Alcoholism (Psychiatric disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 9 | 4
Anxiety disorder (Psychiatric disorders) | 2 | 2
Bipolar I disorder (Psychiatric disorders) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 3 | 1
Confusional state (Psychiatric disorders) | 0 | 2
Delirium (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 14 | 5
Depression suicidal (Psychiatric disorders) | 0 | 2
Disorientation (Psychiatric disorders) | 1 | 0
Drug abuse (Psychiatric disorders) | 0 | 2
Emotional distress (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 0
Major depression (Psychiatric disorders) | 0 | 2
Mental disorder due to a general medical condition (Psychiatric disorders) | 1 | 1
Mental status changes (Psychiatric disorders) | 4 | 5
Mood disorder due to a general medical condition (Psychiatric disorders) | 1 | 0
Psychotic disorder due to a general medical condition (Psychiatric disorders) | 0 | 1
Schizophrenia, undifferentiated type (Psychiatric disorders) | 1 | 0
Substance abuse (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 3
Suicide attempt (Psychiatric disorders) | 1 | 2
Acquired phimosis (Reproductive system and breast disorders) | 1 | 0
Balanoposthitis (Reproductive system and breast disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 12 | 9
Breast pain (Reproductive system and breast disorders) | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0
Cervix disorder (Reproductive system and breast disorders) | 0 | 1
Cystocele (Reproductive system and breast disorders) | 1 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 2 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 1
Organic erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 5 | 2
Perineal fistula (Reproductive system and breast disorders) | 0 | 1
Prostatic disorder (Reproductive system and breast disorders) | 1 | 0
Prostatism (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 3 | 0
Rectocele (Reproductive system and breast disorders) | 1 | 1
Sperm granuloma (Reproductive system and breast disorders) | 1 | 0
Spermatocele (Reproductive system and breast disorders) | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 2
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 3 | 2
Afferent loop syndrome (Injury, poisoning and procedural complications) | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 5
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 3
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 4 | 6
Arterial restenosis (Injury, poisoning and procedural complications) | 2 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 2 | 0
Brain contusion (Injury, poisoning and procedural complications) | 4 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1
Burns third degree (Injury, poisoning and procedural complications) | 1 | 0
Cardiac function disturbance postoperative (Injury, poisoning and procedural complications) | 1 | 1
Cardiac procedure complication (Injury, poisoning and procedural complications) | 2 | 1
Carotid artery restenosis (Injury, poisoning and procedural complications) | 0 | 1
Cerebral hyperperfusion syndrome (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 1 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 3 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 2 | 1
Contrast media reaction (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 5 | 5
Coronary artery reocclusion (Injury, poisoning and procedural complications) | 1 | 0
Coronary artery restenosis (Injury, poisoning and procedural complications) | 30 | 30
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Cystitis radiation (Injury, poisoning and procedural complications) | 0 | 1
Dural tear (Injury, poisoning and procedural complications) | 1 | 0
Electric shock (Injury, poisoning and procedural complications) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Exposure via inhalation (Injury, poisoning and procedural complications) | 0 | 1
Eye penetration (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 3 | 1
Fall (Injury, poisoning and procedural complications) | 6 | 3
Fat embolism (Injury, poisoning and procedural complications) | 0 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 4 | 6
Femur fracture (Injury, poisoning and procedural complications) | 10 | 7
Fibula fracture (Injury, poisoning and procedural complications) | 2 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 3
Foreign body (Injury, poisoning and procedural complications) | 0 | 1
Fractured ischium (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal disorder postoperative (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal injury (Injury, poisoning and procedural complications) | 1 | 0
Graft thrombosis (Injury, poisoning and procedural complications) | 0 | 2
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 2
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 4 | 2
Heart injury (Injury, poisoning and procedural complications) | 0 | 1
Heat exhaustion (Injury, poisoning and procedural complications) | 1 | 0
Heat stroke (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 10 | 11
Humerus fracture (Injury, poisoning and procedural complications) | 5 | 3
Incision site pain (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 2
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 5
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Kidney contusion (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 2 | 2
Ligament rupture (Injury, poisoning and procedural complications) | 2 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 2
Limb injury (Injury, poisoning and procedural complications) | 4 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 3 | 4
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 4
Mountain sickness acute (Injury, poisoning and procedural complications) | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 3 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 1
Overdose (Injury, poisoning and procedural complications) | 4 | 4
Pelvic fracture (Injury, poisoning and procedural complications) | 3 | 1
Peroneal nerve injury (Injury, poisoning and procedural complications) | 1 | 0
Pneumoconiosis (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 4 | 2
Post procedural contusion (Injury, poisoning and procedural complications) | 1 | 0
Post procedural fistula (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 1
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 6 | 3
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 1 | 2
Procedural complication (Injury, poisoning and procedural complications) | 1 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Procedural headache (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0
Pseudomeningocele (Injury, poisoning and procedural complications) | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 3 | 1
Pulmonary contusion (Injury, poisoning and procedural complications) | 2 | 1
Radius fracture (Injury, poisoning and procedural complications) | 2 | 4
Renal haematoma (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 9 | 7
Road traffic accident (Injury, poisoning and procedural complications) | 5 | 3
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1
Scrotal haematoma (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Shunt stenosis (Injury, poisoning and procedural complications) | 2 | 0
Shunt thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Skull fractured base (Injury, poisoning and procedural complications) | 1 | 1
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 3
Splenic injury (Injury, poisoning and procedural complications) | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 2 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 6 | 5
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 2
Tendon injury (Injury, poisoning and procedural complications) | 0 | 2
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 4
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 3 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 4 | 5
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 2
Traumatic shock (Injury, poisoning and procedural complications) | 1 | 0
Traumatic ulcer (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 2
Vascular graft occlusion (Injury, poisoning and procedural complications) | 3 | 0
Vascular graft thrombosis0 (Injury, poisoning and procedural complications) | 0 | 1
Vascular procedure complication (Injury, poisoning and procedural complications) | 0 | 2
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 8 | 2
Wound (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 1
Wound necrosis (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 1
Alanine aminotransferase increased (Investigations) | 4 | 6
Ammonia increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 0 | 1
Blood potassium decreased (Investigations) | 1 | 0
Blood potassium increased (Investigations) | 1 | 1
C-reactive protein increased (Investigations) | 1 | 2
Cardiac enzymes increased (Investigations) | 1 | 1
Cardiac output decreased (Investigations) | 0 | 1
Cardiac stress test abnormal (Investigations) | 1 | 2
Clostridium test positive (Investigations) | 1 | 0
ECG signs of myocardial ischaemia (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 2
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Electrocardiogram ST segment depression (Investigations) | 0 | 2
Electrocardiogram ST segment elevation (Investigations) | 1 | 0
Exercise test abnormal (Investigations) | 3 | 0
Fibrin D dimer increased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 1
Heart rate increased (Investigations) | 1 | 0
Hepatic enzyme abnormal (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 8 | 9
International normalised ratio increased (Investigations) | 0 | 2
Laboratory test abnormal (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Platelet count increased (Investigations) | 0 | 1
Pulmonary function test decreased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Troponin I increased (Investigations) | 1 | 0
Troponin T increased (Investigations) | 1 | 3
Troponin increased (Investigations) | 16 | 7
Weight decreased (Investigations) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 8 | 11
Acute left ventricular failure (Cardiac disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 446 | 432
Angina pectoris (Cardiac disorders) | 272 | 266
Angina unstable (Cardiac disorders) | 546 | 562
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 3 | 2
Arrhythmia (Cardiac disorders) | 3 | 1
Arrhythmia supraventricular (Cardiac disorders) | 1 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 5 | 11
Arteriospasm coronary (Cardiac disorders) | 0 | 3
Atrial fibrillation (Cardiac disorders) | 108 | 76
Atrial flutter (Cardiac disorders) | 14 | 13
Atrial tachycardia (Cardiac disorders) | 0 | 2
Atrial thrombosis (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 2 | 3
Atrioventricular block complete (Cardiac disorders) | 14 | 5
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 4 | 10
Bradyarrhythmia (Cardiac disorders) | 0 | 3
Bradycardia (Cardiac disorders) | 9 | 21
Bundle branch block left (Cardiac disorders) | 2 | 0
Cardiac aneurysm (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 18 | 29
Cardiac asthma (Cardiac disorders) | 2 | 2
Cardiac discomfort (Cardiac disorders) | 1 | 2
Cardiac failure (Cardiac disorders) | 176 | 170
Cardiac failure acute (Cardiac disorders) | 21 | 20
Cardiac failure chronic (Cardiac disorders) | 14 | 16
Cardiac failure congestive (Cardiac disorders) | 101 | 107
Cardiac tamponade (Cardiac disorders) | 2 | 1
Cardio-respiratory arrest (Cardiac disorders) | 9 | 5
Cardiogenic shock (Cardiac disorders) | 5 | 10
Cardiomyopathy (Cardiac disorders) | 1 | 3
Cardiopulmonary failure (Cardiac disorders) | 2 | 1
Cardiorenal syndrome (Cardiac disorders) | 0 | 2
Cardiovascular disorder (Cardiac disorders) | 11 | 10
Cardiovascular insufficiency (Cardiac disorders) | 4 | 1
Chronotropic incompetence (Cardiac disorders) | 1 | 0
Conduction disorder (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 145 | 139
Coronary artery dissection (Cardiac disorders) | 3 | 1
Coronary artery insufficiency (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 10 | 6
Coronary artery perforation (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 59 | 38
Coronary artery thrombosis (Cardiac disorders) | 1 | 0
Dilatation ventricular (Cardiac disorders) | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 1 | 1
Interventricular septum rupture (Cardiac disorders) | 0 | 1
Intracardiac thrombus (Cardiac disorders) | 2 | 3
Ischaemic cardiomyopathy (Cardiac disorders) | 5 | 8
Left ventricular dysfunction (Cardiac disorders) | 1 | 3
Left ventricular failure (Cardiac disorders) | 4 | 6
Microvascular coronary artery disease (Cardiac disorders) | 1 | 0
Mitral valve disease (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 5 | 6
Myocardial fibrosis (Cardiac disorders) | 4 | 1
Myocardial infarction (Cardiac disorders) | 61 | 45
Myocardial ischaemia (Cardiac disorders) | 53 | 47
Myocardial rupture (Cardiac disorders) | 1 | 0
Myopericarditis (Cardiac disorders) | 1 | 0
Nodal rhythm (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 9 | 9
Paroxysmal arrhythmia (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 4 | 2
Pericardial haemorrhage (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 12 | 9
Pleuropericarditis (Cardiac disorders) | 2 | 0
Postinfarction angina (Cardiac disorders) | 8 | 4
Prinzmetal angina (Cardiac disorders) | 1 | 4
Pulseless electrical activity (Cardiac disorders) | 1 | 0
Restrictive cardiomyopathy (Cardiac disorders) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 10 | 7
Sinoatrial block (Cardiac disorders) | 0 | 1
Sinus arrhythmia (Cardiac disorders) | 2 | 1
Sinus bradycardia (Cardiac disorders) | 5 | 3
Sinus tachycardia (Cardiac disorders) | 3 | 0
Stress cardiomyopathy (Cardiac disorders) | 2 | 1
Supraventricular extrasystoles (Cardiac disorders) | 1 | 1
Supraventricular tachyarrhythmia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 11 | 4
Tachyarrhythmia (Cardiac disorders) | 3 | 0
Tachycardia (Cardiac disorders) | 3 | 1
Tachycardia paroxysmal (Cardiac disorders) | 1 | 0
Torsade de pointes (Cardiac disorders) | 1 | 0
Trifascicular block (Cardiac disorders) | 1 | 0
Ventricle rupture (Cardiac disorders) | 2 | 0
Ventricular arrhythmia (Cardiac disorders) | 3 | 4
Ventricular dyssynchrony (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 4 | 5
Ventricular fibrillation (Cardiac disorders) | 14 | 12
Ventricular tachyarrhythmia (Cardiac disorders) | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 28 | 19
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1 | 1
Odontogenic cyst (Congenital, familial and genetic disorders) | 2 | 0
Phimosis (Congenital, familial and genetic disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 16 | 9
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 | 7
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Asthma late onset (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 45 | 56
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 27 | 21
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 | 6
Granulomatous pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 | 14
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 9 | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 22 | 28
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 18 | 15
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11 | 11
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 43 | 49
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 1
Aplastic anaemia (Blood and lymphatic system disorders) | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 3 | 3
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Hypercoagulation (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 7 | 6
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 | 0
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 2 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2
Aphasia (Nervous system disorders) | 2 | 1
Ataxia (Nervous system disorders) | 0 | 2
Basilar migraine (Nervous system disorders) | 1 | 0
Brain injury (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 2 | 1
Brain stem stroke (Nervous system disorders) | 0 | 3
Carotid arteriosclerosis (Nervous system disorders) | 3 | 3
Carotid artery disease (Nervous system disorders) | 1 | 5
Carotid artery occlusion (Nervous system disorders) | 2 | 0
Carotid artery stenosis (Nervous system disorders) | 34 | 27
Carotid sinus syndrome (Nervous system disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 3 | 0
Cerebellar ataxia (Nervous system disorders) | 1 | 0
Cerebellar haemorrhage (Blood and lymphatic system disorders) | 1 | 1
Cerebellar infarction (Nervous system disorders) | 1 | 1
Cerebral arteriosclerosis (Nervous system disorders) | 2 | 0
Cerebral artery embolism (Nervous system disorders) | 0 | 1
Cerebral circulatory failure (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 2 | 7
Cerebral infarction (Nervous system disorders) | 6 | 3
Cerebral ischaemia (Nervous system disorders) | 3 | 4
Cerebrovascular accident (Nervous system disorders) | 16 | 19
Cerebrovascular disorder (Nervous system disorders) | 0 | 1
Cerebrovascular insufficiency (Nervous system disorders) | 1 | 0
Cervical myelopathy (Nervous system disorders) | 1 | 0
Cervical neuritis (Nervous system disorders) | 0 | 1
Cervical radiculopathy (Nervous system disorders) | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | 2 | 2
Cognitive disorder (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 3 | 1
Complex regional pain syndrome (Nervous system disorders) | 0 | 3
Convulsion (Nervous system disorders) | 8 | 6
Dementia (Nervous system disorders) | 1 | 1
Dementia Alzheimer's type (Nervous system disorders) | 0 | 2
Diabetic neuropathy (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 7 | 13
Dysaesthesia (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 1
Embolic stroke (Nervous system disorders) | 4 | 4
Encephalopathy (Nervous system disorders) | 0 | 2
Epilepsy (Nervous system disorders) | 3 | 4
Frontotemporal dementia (Nervous system disorders) | 1 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 2
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 | 2
Haemorrhagic stroke (Nervous system disorders) | 10 | 6
Haemorrhagic transformation stroke (Nervous system disorders) | 3 | 1
Head discomfort (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 4 | 4
Hemiparesis (Nervous system disorders) | 1 | 0
Hemiplegia (Nervous system disorders) | 1 | 0
Hemiplegic migraine (Nervous system disorders) | 1 | 1
Hyperaesthesia (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 5 | 3
Hypoglycaemic coma (Nervous system disorders) | 0 | 1
Hypoglycaemic seizure (Nervous system disorders) | 0 | 1
Hypotonia (Nervous system disorders) | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 1
Intercostal neuralgia (Nervous system disorders) | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 2 | 0
Intracranial haematoma (Nervous system disorders) | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 9 | 14
Ischaemic stroke (Nervous system disorders) | 86 | 93
Lacunar infarction (Nervous system disorders) | 4 | 3
Lethargy (Nervous system disorders) | 1 | 3
Loss of consciousness (Nervous system disorders) | 3 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 2
Monoparesis (Nervous system disorders) | 1 | 0
Monoplegia (Nervous system disorders) | 1 | 0
Motor neurone disease (Nervous system disorders) | 0 | 1
Multiple sclerosis relapse (Nervous system disorders) | 1 | 0
Narcolepsy (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 1
Neuroglycopenia (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 2
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 1
Occipital neuralgia (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 2 | 3
Paraplegia (Nervous system disorders) | 0 | 1
Paresis (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Postictal paralysis (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 12 | 9
Radiculopathy (Nervous system disorders) | 1 | 2
Sciatica (Nervous system disorders) | 4 | 5
Sensory disturbance (Nervous system disorders) | 0 | 1
Simple partial seizures (Nervous system disorders) | 1 | 0
Speech disorder (Nervous system disorders) | 1 | 0
Spinal epidural haematoma (Nervous system disorders) | 0 | 1
Spondylitic myelopathy (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 10 | 5
Syncope (Nervous system disorders) | 60 | 58
Thalamic infarction (Nervous system disorders) | 0 | 1
Transient global amnesia (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 45 | 48
Trigeminal neuralgia (Nervous system disorders) | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 1 | 0
Vascular encephalopathy (Nervous system disorders) | 0 | 1
Vertebral artery occlusion (Nervous system disorders) | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 6 | 1
Vertigo CNS origin (Nervous system disorders) | 0 | 1
Accommodation disorder (Eye disorders) | 0 | 1
Age-related macular degeneration (Eye disorders) | 0 | 1
Amaurosis fugax (Eye disorders) | 1 | 1
Blindness (Eye disorders) | 1 | 0
Blindness unilateral (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 4 | 12
Cataract nuclear (Eye disorders) | 0 | 1
Diabetic retinopathy (Eye disorders) | 0 | 1
Diplopia (Nervous system disorders) | 1 | 0
Ectropion (Nervous system disorders) | 0 | 1
Eye haemorrhage (Eye disorders) | 1 | 2
Eyelid cyst (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 0 | 1
Lens dislocation (Eye disorders) | 0 | 1
Macular hole (Eye disorders) | 1 | 0
Open angle glaucoma (Eye disorders) | 1 | 0
Optic neuropathy (Eye disorders) | 0 | 1
Retinal artery occlusion (Eye disorders) | 1 | 1
Retinal detachment (Eye disorders) | 2 | 3
Retinal haemorrhage (Eye disorders) | 2 | 0
Retinoschisis (Eye disorders) | 0 | 1
Visual acuity reduced (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 2
Deafness (Ear and labyrinth disorders) | 0 | 1
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 2 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 8 | 8
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Vestibular disorder (Ear and labyrinth disorders) | 1 | 1
Abdominal adhesions (Gastrointestinal disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 6
Abdominal pain (Gastrointestinal disorders) | 12 | 8
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 9 | 8
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0
Abnormal faeces (Gastrointestinal disorders) | 1 | 0
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 3 | 0
Anal fistula (Gastrointestinal disorders) | 2 | 3
Barrett's oesophagus (Gastrointestinal disorders) | 1 | 0
Brunner's gland hyperplasia (Gastrointestinal disorders) | 1 | 0
Caecitis (Gastrointestinal disorders) | 0 | 1
Coeliac artery stenosis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 5
Colitis ischaemic (Gastrointestinal disorders) | 2 | 2
Colitis ulcerative (Gastrointestinal disorders) | 1 | 1
Colonic pseudo-obstruction (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 6
Crohn's disease (Gastrointestinal disorders) | 1 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 1 | 0
Diaphragmatic hernia (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 14
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 8
Diverticulum intestinal (Gastrointestinal disorders) | 5 | 4
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1
Duodenal polyp (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 7 | 5
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 3 | 2
Duodenitis (Gastrointestinal disorders) | 1 | 2
Duodenogastric reflux (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 5 | 7
Dysphagia (Gastrointestinal disorders) | 2 | 0
Enteritis (Gastrointestinal disorders) | 1 | 1
Enterocele (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 2 | 1
Enterovesical fistula (Gastrointestinal disorders) | 2 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 2
Faeces discoloured (Gastrointestinal disorders) | 0 | 1
Femoral hernia (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 4
Gastric haemorrhage (Gastrointestinal disorders) | 5 | 2
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 2 | 0
Gastric ulcer (Gastrointestinal disorders) | 17 | 13
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 | 2
Gastritis (Gastrointestinal disorders) | 16 | 10
Gastritis atrophic (Gastrointestinal disorders) | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 3 | 3
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 1
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastroduodenitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 3 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 26 | 18
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 13 | 6
Gastrooesophagitis (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 3 | 3
Haematochezia (Gastrointestinal disorders) | 1 | 1
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 | 2
Haemorrhoids (Gastrointestinal disorders) | 3 | 2
Hiatus hernia (Gastrointestinal disorders) | 4 | 5
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 1
Ileal perforation (Gastrointestinal disorders) | 1 | 0
Ileal stenosis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 3 | 3
Ileus paralytic (Gastrointestinal disorders) | 1 | 2
Inguinal hernia (Gastrointestinal disorders) | 17 | 16
Inguinal hernia, obstructive (Gastrointestinal disorders) | 2 | 2
Intestinal haemorrhage (Gastrointestinal disorders) | 2 | 2
Intestinal infarction (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 3 | 2
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Intestinal ulcer (Gastrointestinal disorders) | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 2
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Large intestinal ulcer (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 2
Large intestine polyp (Gastrointestinal disorders) | 8 | 7
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 5
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 2
Megacolon (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 2 | 4
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 6 | 5
Obstruction gastric (Gastrointestinal disorders) | 1 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 1
Oesophageal disorder (Gastrointestinal disorders) | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 2 | 0
Oesophagitis (Gastrointestinal disorders) | 2 | 2
Pancreatic disorder (Gastrointestinal disorders) | 0 | 1
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 7 | 4
Pancreatitis acute (Gastrointestinal disorders) | 11 | 12
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0
Pancreatitis relapsing (Gastrointestinal disorders) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 2 | 1
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Peptic ulcer perforation (Gastrointestinal disorders) | 1 | 0
Periproctitis (Gastrointestinal disorders) | 1 | 0
Peritoneal adhesions (Gastrointestinal disorders) | 1 | 0
Peritoneal mesothelial hyperplasia (Gastrointestinal disorders) | 1 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 1 | 1
Radicular cyst (Gastrointestinal disorders) | 1 | 0
Rectal fissure (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 9 | 7
Rectal polyp (Gastrointestinal disorders) | 0 | 2
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Reflux gastritis (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 5
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 1
Short-bowel syndrome (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 7 | 0
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Small intestine polyp (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 2 | 2
Umbilical hernia (Gastrointestinal disorders) | 3 | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 8 | 10
Uraemic gastropathy (Gastrointestinal disorders) | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 6 | 4
Metrorrhagia (Reproductive system and breast disorders) | 2 | 0
Acute prerenal failure (Renal and urinary disorders) | 2 | 0
Azotaemia (Renal and urinary disorders) | 1 | 1
Bladder outlet obstruction (Renal and urinary disorders) | 1 | 1
Bladder stenosis (Renal and urinary disorders) | 1 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 3
Calculus ureteric (Renal and urinary disorders) | 2 | 4
Calculus urethral (Renal and urinary disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 3 | 3
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 13 | 9
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 2
Hydronephrosis (Renal and urinary disorders) | 1 | 1
Hypertensive nephropathy (Renal and urinary disorders) | 0 | 1
Micturition disorder (Renal and urinary disorders) | 0 | 1
Nephritis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 9 | 8
Nephropathy (Renal and urinary disorders) | 0 | 2
Nephrotic syndrome (Renal and urinary disorders) | 3 | 0
Polyuria (Renal and urinary disorders) | 0 | 1
Renal artery arteriosclerosis (Renal and urinary disorders) | 0 | 1
Renal artery occlusion (Renal and urinary disorders) | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 3 | 6
Renal colic (Renal and urinary disorders) | 2 | 6
Renal failure (Renal and urinary disorders) | 19 | 20
Renal failure acute (Renal and urinary disorders) | 46 | 44
Renal failure chronic (Renal and urinary disorders) | 5 | 16
Renal haemorrhage (Renal and urinary disorders) | 1 | 0
Renal hypertension (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 5 | 7
Renal infarct (Renal and urinary disorders) | 2 | 0
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0
Ureteric dilatation (Renal and urinary disorders) | 0 | 1
Ureteric haemorrhage (Renal and urinary disorders) | 1 | 0
Urethral haemorrhage (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 2 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0
Urinary bladder polyp (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 8 | 1
Urinoma (Renal and urinary disorders) | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 0 | 2
Alcoholic liver disease (Hepatobiliary disorders) | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 2 | 0
Bile duct obstruction (Hepatobiliary disorders) | 2 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 2
Bile duct stone (Hepatobiliary disorders) | 3 | 4
Biliary colic (Hepatobiliary disorders) | 1 | 2
Biliary dyskinesia (Hepatobiliary disorders) | 2 | 0
Cholangitis (Hepatobiliary disorders) | 3 | 2
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 13 | 10
Cholecystitis acute (Hepatobiliary disorders) | 15 | 15
Cholecystitis chronic (Hepatobiliary disorders) | 3 | 0
Cholelithiasis (Hepatobiliary disorders) | 18 | 23
Cholestasis (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 3 | 7
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatic cyst (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 4
Hepatic function abnormal (Hepatobiliary disorders) | 5 | 2
Hepatitis (Hepatobiliary disorders) | 3 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Hepatitis alcoholic (Hepatobiliary disorders) | 1 | 0
Hepatitis cholestatic (Hepatobiliary disorders) | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 1 | 1
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 2 | 0
Hepatotoxicity (Hepatobiliary disorders) | 2 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 3 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 8 | 2
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Dry gangrene (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Pemphigus (Skin and subcutaneous tissue disorders) | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 7 | 9
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 6 | 7
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 8
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Fracture malunion (Musculoskeletal and connective tissue disorders) | 0 | 1
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 2 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 11 | 9
Joint instability (Musculoskeletal and connective tissue disorders) | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 4
Muscle disorder (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 21 | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 3
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 40 | 29
Osteochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 6
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Plantar fascial fibromatosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1
Polymyositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 3 | 7
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 2
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 | 6
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 9
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 3 | 1
Spondylolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Sympathetic posterior cervical syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Autoimmune thyroiditis (Endocrine disorders) | 0 | 2
Goitre (Endocrine disorders) | 4 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 2
Primary hypothyroidism (Endocrine disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 18 | 19
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 19 | 17
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 | 4
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 3 | 1
Hydraemia (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 6
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 11 | 13
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 10 | 6
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 2 | 3
Insulin-requiring type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 2 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 21 | 21
Abdominal abscess (Infections and infestations) | 1 | 1
Abdominal infection (Infections and infestations) | 1 | 0
Abdominal wall abscess (Metabolism and nutrition disorders) | 3 | 0
Abscess (Infections and infestations) | 2 | 1
Abscess intestinal (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 6 | 2
Acarodermatitis (Infections and infestations) | 0 | 1
Acute tonsillitis (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 6 | 3
Appendiceal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 8 | 9
Appendicitis perforated (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 3
Arthritis infective (Infections and infestations) | 2 | 0
Bacteraemia (Infections and infestations) | 2 | 0
Bacterial prostatitis (Infections and infestations) | 0 | 1
Bone abscess (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 19 | 29
Bronchopneumonia (Infections and infestations) | 10 | 9
Burkholderia pseudomallei infection (Infections and infestations) | 0 | 2
Bursitis infective (Infections and infestations) | 0 | 1
Campylobacter infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 24 | 27
Cellulitis staphylococcal (Infections and infestations) | 2 | 0
Cholangitis suppurative (Infections and infestations) | 1 | 1
Cholecystitis infective (Infections and infestations) | 2 | 1
Chronic sinusitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 5 | 3
Clostridium difficile infection (Infections and infestations) | 7 | 2
Creutzfeldt-Jakob disease (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 6 | 2
Cytomegalovirus infection (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 2 | 1
Device related sepsis (Infections and infestations) | 1 | 0
Diabetic foot infection (Infections and infestations) | 1 | 1
Diabetic gangrene (Infections and infestations) | 1 | 2
Diarrhoea infectious (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 16 | 14
Eczema infected (Infections and infestations) | 0 | 1
Empyema (Infections and infestations) | 2 | 0
Endocarditis (Infections and infestations) | 2 | 1
Endocarditis enterococcal (Infections and infestations) | 1 | 0
Enteritis infectious (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 2
Erysipelas (Infections and infestations) | 4 | 6
Escherichia urinary tract infection (Infections and infestations) | 3 | 1
Gallbladder abscess (Infections and infestations) | 0 | 1
Gallbladder empyema (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 8 | 7
Gastric infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 20 | 18
Gastroenteritis clostridial (Infections and infestations) | 2 | 0
Gastroenteritis norovirus (Infections and infestations) | 2 | 0
Gastroenteritis viral (Infections and infestations) | 2 | 2
Gastrointestinal infection (Infections and infestations) | 1 | 1
Graft infection (Infections and infestations) | 1 | 1
Groin abscess (Infections and infestations) | 2 | 0
Groin infection (Infections and infestations) | 2 | 0
Haematoma infection (Infections and infestations) | 1 | 1
Helicobacter infection (Infections and infestations) | 1 | 0
Hepatitis C (Infections and infestations) | 2 | 1
Hepatitis E (Infections and infestations) | 1 | 0
Hepatitis infectious mononucleosis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 3 | 1
Impetigo (Infections and infestations) | 0 | 1
Infected dermal cyst (Infections and infestations) | 1 | 0
Infected lymphocele (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 4 | 2
Infection (Infections and infestations) | 1 | 2
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 2 | 1
Influenza (Infections and infestations) | 4 | 3
Klebsiella infection (Infections and infestations) | 1 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 1
Labyrinthitis (Infections and infestations) | 2 | 2
Liver abscess (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 4 | 4
Localised infection (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 4
Lung abscess (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 2 | 3
Lymphangitis (Infections and infestations) | 0 | 1
Malaria (Infections and infestations) | 1 | 1
Mastoiditis (Infections and infestations) | 0 | 2
Mediastinitis (Infections and infestations) | 1 | 0
Meningitis tuberculous (Infections and infestations) | 1 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 2
Neuroborreliosis (Infections and infestations) | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 1 | 2
Osteomyelitis (Infections and infestations) | 2 | 7
Osteomyelitis acute (Infections and infestations) | 1 | 0
Osteomyelitis chronic (Infections and infestations) | 1 | 2
Otitis media (Infections and infestations) | 1 | 0
Pelvic abscess (Infections and infestations) | 1 | 0
Pericarditis tuberculous (Infections and infestations) | 1 | 0
Peritoneal abscess (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 2 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 113 | 130
Pneumonia bacterial (Infections and infestations) | 2 | 1
Pneumonia fungal (Infections and infestations) | 1 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 1
Pneumonia pseudomonas aeruginosa (Infections and infestations) | 0 | 2
Pneumonia staphylococcal (Infections and infestations) | 1 | 1
Pneumonia streptococcal (Infections and infestations) | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 3
Post procedural pneumonia (Infections and infestations) | 0 | 1
Post procedural sepsis (Infections and infestations) | 0 | 1
Postoperative abscess (Infections and infestations) | 2 | 0
Postoperative wound infection (Infections and infestations) | 4 | 6
Pseudomembranous colitis (Infections and infestations) | 2 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 2
Pulmonary tuberculosis (Infections and infestations) | 1 | 1
Pyelonephritis (Infections and infestations) | 5 | 3
Pyelonephritis acute (Infections and infestations) | 4 | 1
Pyoderma streptococcal (Infections and infestations) | 0 | 1
Renal abscess (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 5 | 5
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Salmonellosis (Infections and infestations) | 2 | 0
Scrotal abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 23 | 24
Septic shock (Infections and infestations) | 9 | 6
Sinusitis (Infections and infestations) | 2 | 3
Skin bacterial infection (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal abscess (Infections and infestations) | 0 | 2
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 3
Staphylococcal sepsis (Infections and infestations) | 3 | 1
Staphylococcal skin infection (Infections and infestations) | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 2
Subcutaneous abscess (Infections and infestations) | 1 | 1
Superinfection (Infections and infestations) | 0 | 1
Testicular abscess (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 6 | 5
Upper respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 47 | 25
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Urinary tract infection enterococcal (Infections and infestations) | 2 | 0
Urinary tract infection pseudomonal (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 6 | 7
Vestibular neuronitis (Infections and infestations) | 2 | 1
Viral infection (Infections and infestations) | 4 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 5 | 5
Wound infection pseudomonas (Infections and infestations) | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 0 | 1
Wound sepsis (Infections and infestations) | 0 | 2
Pneumonia legionella (Infections and infestations) | 0 | 1
Cerebellar haemorrhage (Nervous system disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6465) | Darapladib 160 mg (N=6452)
Hypertension (Vascular disorders) | 409 | 370
Hypotension (Vascular disorders) | 132 | 154
Angina pectoris (Cardiac disorders) | 398 | 363
Atrial fibrillation (Cardiac disorders) | 185 | 154
Cough (Respiratory, thoracic and mediastinal disorders) | 355 | 324
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 310 | 286
Anaemia (Blood and lymphatic system disorders) | 187 | 184
Dizziness (Nervous system disorders) | 357 | 354
Headache (Nervous system disorders) | 202 | 175
Chest discomfort (General disorders) | 111 | 134
Fatigue (General disorders) | 334 | 302
Non-cardiac chest pain (General disorders) | 431 | 414
Oedema peripheral (General disorders) | 245 | 239
Abdominal pain (Gastrointestinal disorders) | 130 | 140
Abdominal pain upper (Gastrointestinal disorders) | 128 | 135
Abnormal faeces (Gastrointestinal disorders) | 64 | 525
Constipation (Gastrointestinal disorders) | 174 | 165
Diarrhoea (Gastrointestinal disorders) | 351 | 675
Dyspepsia (Gastrointestinal disorders) | 116 | 130
Large intestine polyp (Gastrointestinal disorders) | 130 | 127
Nausea (Gastrointestinal disorders) | 176 | 198
Urine odour abnormal (Renal and urinary disorders) | 65 | 344
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 23 | 241
Arthralgia (Musculoskeletal and connective tissue disorders) | 207 | 158
Back pain (Musculoskeletal and connective tissue disorders) | 262 | 224
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 130 | 98
Myalgia (Musculoskeletal and connective tissue disorders) | 186 | 215
Pain in extremity (Musculoskeletal and connective tissue disorders) | 221 | 181
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 358 | 325
Bronchitis (Infections and infestations) | 178 | 192
Influenza (Infections and infestations) | 143 | 141
Nasopharyngitis (Infections and infestations) | 279 | 273
Upper respiratory tract infection (Infections and infestations) | 144 | 162
Urinary tract infection (Infections and infestations) | 205 | 157

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.